CLINICAL TRIAL: NCT03775044
Title: Assessment of Medherent Medication Management Device and Adherence Platform
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terrapin Pharmacy (Industry)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Joel F. Feldman, President, Terrapin Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R44MH116765-01 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Mental Health Disorder; Medication Adherence
Keywords: Telemedicine; Medication Adherence; Mental Health Issue
MeSH Terms: conditions — Mental Disorders; Medication Adherence

STUDY DESIGN:
Intervention Model Description: This study is a stepped wedge design where all individuals receive the intervention but at different time points after enrollment in the study. Each person will have two observations before the intervention and three observations after the intervention. Health service use data will be collected for two years prior to enrollment and two years after enrollment.
Masking Description: No masking is possible for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: Medherent Device (Experimental): All participants get the Medherent device. There is only one arm to this study.
  Interventions: Device: Medherent Device

INTERVENTIONS:
Device: Medherent Device — The Medherent Medication Management Device (MMD) is intended to enable patients to self-manage their medication at home when it may otherwise require assistance.

SUMMARY:
This study uses a stepped wedge designs to estimate the effect of using the Medherent Medication Management Device on medication adherence for a population of 150 individuals who are diagnosed with serious mental illness.

DETAILED DESCRIPTION:
Individuals suffering from Serious Mental Illnesses (SMI) such as schizophrenia, bipolar disorder or depressive disorders are at risk for serious adverse psychiatric, other health, and social outcomes. Essential to controlling chronic psychiatric and health disorders is adherence to medications that are prescribed to address the symptoms and causes of these health conditions. Medication adherence is particularly challenging for those with SMI. Good adherence is defined as 80% or more of medication taken, whereas the average patient with schizophrenia or bipolar disorder takes 50-70% of prescribed medications. For individuals with SMI, important barriers to adherence include cognitive impairments and lack of illness insight, meaning that they are not aware of the symptoms and consequences of their illness. Inquiries about drug intake by psychiatrists, relatives, or others has been linked to greater adherence. Positive relationships with physicians, psychiatrists and their staff have been found to be significant predictors of good adherence in SMI patients, while difficulties in building a therapeutic alliance and poor clinical-patient relationship are significant predictors of nonadherence. Failure to recognize nonadherence may prompt physicians to misattribute poor outcomes to treatment failure, leading to inappropriate dosage increases or unnecessary medication switches. Moreover, non- adherence in SMI patients is associated with greater economic and social burden, due to higher hospitalization rates, longer hospital stays, more emergency room and emergency psychiatric visits, greater risk of suicide and violence towards others, and higher rates of deleterious psychotic relapses.

The Medherent© Medication Management Device (MMD) is a tool developed by Terrapin Pharmacy to improve medication adherence through the integration of medication dispensing and prompts to consumers to take medications, with real-time electronic feedback to care managers about consumers' adherence behaviors and daily health status. This MMD builds on adherence interventions proven effective in SMI patients and enables care managers to expand the number of individuals that they can care for effectively.

This study uses a stepped-wedge design with 150 individuals across all study sites and approximately 150 individuals to answer the following aims:

1. Measure the effect of the Medherent platform and interventions on adherence and medication use.

   1. Measure change in adherence by triangulating self-report data, clinician observation, biological measures, chart reviews and clinical outcomes before and after exposure to the Medherent intervention. Medherent device data will also be used to measure the consumer levels of adherence to medications.
   2. Document pharmacy interaction issues (e.g. arranging refill times, responsiveness to prescription changes), device fail rate, and remaining user interface issues (e.g. acceptability of adherence prompts, operating system issues).
2. Measure the effect of Medherent use on clinical outcomes and health service costs.

   1. Change in clinical relationships, attitudes about medications, and acute care service use (e.g. hospitalizations and emergency department visits) will be measured by consumer interviews, chart reviews, Medherent dispensing data, and claims data (Medicaid)
   2. Using Medicaid data, pharmacy data, and agency clinical data we will develop a cost model for Medherent users before and after enrollment and develop a matched comparison group using other Maryland Medicaid recipients who have not been enrolled in the Medherent treatment arm to measure changes in health service utilization and the corresponding costs.

ELIGIBILITY:
Inclusion Criteria:

* Currently be a client of a participating community mental health agency
* Have a diagnoses mental illness
* Currently be prescribed a psychotropic medication for the purpose of treatment a mental illness
* Be able to consent to participants in the study
* Be over 18 years old and under 80 years old

Exclusion Criteria:

* Under 18 years old.
* Over 80 years old.
* Unable to consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Evaluation of Medication Influences and Beliefs (BEMIB) Adherence Measure | Change between enrollment/baseline and follow up measures (1 month, 6 month, 12 month)
  Brief Evaluation of Medication Influences and Beliefs (BEMIB) is an 8-item scale. Total scores range from 0 to 32 with higher scores indicating more negative beliefs about medications.
Voils two-part measure of medication nonadherence | Change between enrollment/baseline and follow up measures (1 month, 6 month, 12 month)
  Measure of extent of non adherence and reasons for non-adherence The extent of non-adherence scale averages scores over the 3 items and range from 1-5. The measure is continuous with higher scores indicating higher adherence. The reasons for non adherence scale is comprised of 24 reasons for non adherence and are scored individually from 1 to 5 with higher scores indicating more reasons for non adherence.
Change in Medication Records | Change between weekly adherence from enrollment/baseline compared with weekly adherence for the year after receiving the Medherent Machine
  Chart reviews for medication dispensing records and device dispensing data. Data will be combined to create a variable of medication taking behaviors. If an individual had a recorded dose received/dispensed they will be considered to have taken the dose if a dose was not received/dispensed they will be considered to have not taken a dose. Above 80% doses per week will be considered high adherence, 70-79% medium adherence and below 70% low adherence.
Chart review of clinical records for change in level of adherence support | Change level of adherence support from enrollment/baseline compared to adherence support for the year after receiving the Medherent Machine (e.g. Treatment)
  Level of staff medication support including categories. High Support = Mandatory daily supervision, Medium Support = pill count, low support = self-monitoring of medications
Pharmacy interaction outcomes: Refill Times | Data will be measured continuously for 1 year after receiving the Medherent Machine (e.g. Treatment)
  Counts of days with out prescribed medication including days missed due to missed refills or gaps between receipt of prescription changes at the pharmacy till medication is refilled.
Pharmacy interaction outcomes: Medherent device fail/error rate | Data will be measured continuously for 1 year after receiving the Medherent Machine (e.g. Treatment)
  Counts of device failures or user interface issues that cause a missed dose. Counts will be of missed doses per installed device

SECONDARY OUTCOMES:
Psychiatric Acute Events | Measured from two years prior to Medherent device installation through 1 year after device installation.
  Record of psychiatric acute events
Costs of Services | Measured from two years prior to Medherent device installation through 1 year after device installation.
  Medicaid and mental health agency costs data for calculating the cost of service.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Feldman, JD, Principal Investigator — Terrapin Pharmacy
Locations (1):
- Terrapin Pharmacy, Annapolis, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De identified participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: Four years after the completion of the study.
Access Criteria: We will make the data and associated documentation available to investigators who are working under an institution with a Federal Wide Assurance (FWA) and who agree to a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) appropriate Intuitional Review Board approval for data use; (3) a commitment to securing the data using appropriate computer technology; and (4) a commitment to destroying or returning the data after analyses are completed.